CLINICAL TRIAL: NCT05424029
Title: Extracellular Vesicles and Particles (EVP) as Biomarkers of Recurrence in Non-Small Cell Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 22-155
Record Dates: First submitted 2022-06-14; First posted 2022-06-21 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Extracellular Vesicles and Particles; Biomarkers; 22-155
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — bronchial washings
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to find out if fluid rinsed from peoples' airways (bronchial washing samples) during routine surgery to remove (resect) their non-small cell lung cancer (NSCLC) tumors contains enough vesicles to do testing that may help the researchers learn more about their NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* All patients ≥ 18 years of age undergoing consideration of surgical resection, including lobar resections, sublobar resections, and pneumonectomies, for primary lung cancer will be eligible.
* Patients with previously resected disease and/or previous radiation therapy will be considered on a case by case basis.

Exclusion Criteria:

* Patients with active infection or pneumonia which may impact exosome makeup
* Additionally, if at the discretion of the operating surgeon, obtaining bronchial washings would lead to undue morbidity, the patient would be excluded and replaced

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A member of the patient's treatment team, the protocol investigator, or the research team at MSK will identify potential research subjects
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-06-14 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
to isolate exosomes from bronchial washings | day 1
  every patient from whom the essential specimens have been acquired will be evaluated to determine if more than 100,000 microvesicles can be isolated for exosome purification

CONTACTS AND LOCATIONS:
Overall Officials: David Jones, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Consent Only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent Only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent Only), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Consent Only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent Only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Consent Only), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm